CLINICAL TRIAL: NCT06281834
Title: Dolutegravir Pharmacokinetics During Weekly Rifapentine/Isoniazid for TB Prevention
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: APIN Public Health Initiatives (Unknown); University of Cape Town (Other)
Responsible Party: Principal Investigator, Holly Rawizza, M.D., M.P.H., Assistant Professor of Medicine, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024P000306
Record Dates: First submitted 2024-02-16; First posted 2024-02-28 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Pediatric HIV Infection; Latent Tuberculosis
Keywords: Pediatric HIV; rifapentine; TB prevention
MeSH Terms: conditions — Latent Tuberculosis | interventions — rifapentine; dolutegravir

STUDY DESIGN:
Intervention Model Description: Prospective single-arm, open-label, pharmacokinetic and safety study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dolutegravir PK during weekly rifapentine/isoniazid for TB prevention (Experimental): This is a single arm study: all patients are started on standard HIV treatment, with LTBI/TB prevention treatment varying according to age cohorts. Children 2-11 years receive standard weekly rifapentine/isoniazid (3HP) for TB prevention; those <2 years received a single-dose of extrapolated weekly RPT/INH, followed by standard INH prophylaxis.
  Interventions: Drug: Rifapentine; Drug: Dolutegravir

INTERVENTIONS:
Drug: Rifapentine — Children 2-11 years received standard HIV treatment and 3HP (RPT/INH weekly for 12 weeks) for TB prevention. Children <2 years receive standard HIV treatment, a single-dose of extrapolated weekly RPT/INH, followed by standard INH prophylaxis. Safety and pharmacokinetics will be evaluated.
Drug: Dolutegravir — All children in this study are living with HIV and thus dolutegravir is a standard part of treatment; in this study we will collect blood samples to measure dolutegravir levels during combination treatment with rifapentine/isoniazid treatment for TB prevention

SUMMARY:
Tuberculosis (TB) is the leading cause of death among children living with HIV, yet insufficient data are available on the pharmacokinetics of newer TB prevention strategies in children. Short-course TB prevention/latent TB infection (LTBI) treatment regimens increase completion rates but have not been adequately studied among children living with HIV. Our prospective, open-label PK study will examine and extend use of weekly rifapentine and isoniazid (3HP) among children receiving dolutegravir. This will address gaps in knowledge by examining two-way PK of short-course LTBI treatment in a vulnerable pediatric population.

DETAILED DESCRIPTION:
This study is a prospective, single-arm, open-label, intensive and sparse pharmacokinetic (PK) and safety study to evaluate steady-state dolutegravir (DTG) and rifapentine (RPT) concentrations among 25 ART-naïve or experienced children living with HIV who screen negative for TB in two age categories. Study design differs by age cohort since RPT dosing is well-established for children ≥2 years of age but not for children <2 years. Children 2-11 years receive standard weekly rifapentine/isoniazid (3HP) dosing for a 12-week course, a World Health Organization (WHO)-recommended LTBI treatment option. For young children <2 years of age, intensive PK will be evaluated after a single-dose of extrapolated weekly rifapentine/isoniazid (RPT/INH), followed by standard WHO-recommended LTBI prophylaxis (isoniazid daily).

Children will be recruited from two large pediatric HIV clinics in Nigeria. Children 2-11 years will receive HIV treatment that is considered standard of care consisting of weight-based DTG once daily along with two non-nucleoside reverse transcriptase inhibitors (NRTIs), plus 3HP at standard doses for LTBI treatment. Children <2 years of age also receive standard DTG-based ART as well as standard isoniazid (INH) prophylaxis for LTBI, however, they will additionally receive a single dose of weekly RPT/INH for study purposes. The primary study intervention is, therefore, additional blood sampling for drug concentration determination (both DTG and RPT) and biomarker assessment. Clinical and laboratory monitoring for toxicity occur throughout the 48 week study period.

PK sampling for drug concentration determination will occur at three time points during the 48-week study. Specifically, intensive PK sampling will occur at study week 6, while sparse PK sampling will occur at weeks 4 and 7. Additionally, the endogenous biomarker of CYP3A4 activity, 4-beta-hydroxycholesterol to cholesterol ratio, will be evaluated to advance understanding of underlying mechanisms of drug action. Blood sampling to quantify this biomarker will occur at either 4 (among ART-experienced children) or 5 (ART-naive) time points during the 48-week study.

ELIGIBILITY:
Inclusion Criteria:

* (1) ART-naïve or ART-experienced HIV-infected children 4 weeks to <12 years of age;
* (2) no evidence of active TB based on an appropriate clinical evaluation;
* (3) negative TB diagnostic test if performed (other than tuberculin skin testing);
* (4) weight of at least 4 kilograms; and
* (5) consent of the parent or legal guardian and assent of the child (if ≥7 years of age).

Exclusion Criteria:

* (1) Baseline labs with evidence of ≥grade 3 abnormalities: alanine aminotransferase (ALT), total bilirubin, absolute neutrophil count (ANC), platelets, creatinine;
* (2) presenting with acute respiratory distress or decompensation, or any clinical syndrome which could suggest undiagnosed TB or other opportunistic infection; or
* (3) receipt of a medication that has drug-drug interactions with DTG or RPT.

Ages: 4 Weeks to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Dolutegravir AUC during weekly rifapentine/isoniazid | Weeks 4 and 6
  Dolutegravir area under the concentration time curve (AUC) will be compared to therapeutic ranges established in the adult and pediatric literature. Intensive PK sampling will occur at week 6 for dolutegravir and rifapentine PK. Week 4 sparse PK sampling will provide dolutegravir exposures without rifapentine.

SECONDARY OUTCOMES:
Rifapentine AUC | weeks 6 and 7
  Rifapentine AUC will be compared against adult targets. Week 7 sparse PK will provide weekly Cmin estimate.
Proportion of participants experiencing severe (grade 3 or 4) clinical or laboratory adverse events | Week 48
  Laboratory and clinical toxicities are monitored at 8-9 time points throughout the study and the proportion of children experiencing severe adverse events will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Holly Rawizza, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- University College Hospital, Ibadan, Oyo State, Nigeria

IPD SHARING:
Plan to Share IPD: Yes
At the request of researchers de-identified data may be shared.
Supporting Information: Study Protocol, CSR
Time Frame: After all data are analyzed and results are published.
Access Criteria: At the request of researchers de-identified data may be shared.